CLINICAL TRIAL: NCT06960343
Title: Long Term Clinical Outcome After Arthroscopic Rotator Cuff Repair Augmentation With Autologous Microfragmented Lipoaspirate Tissue: a Prospective Randomized Controlled Trialin Question Won by Our Research Group.
Brief Title: Long Term Clinical Outcome After Arthroscopic Rotator Cuff Repair Augmentation With Autologous Microfragmented Lipoaspirate Tissue
Status: Recruiting | Type: Observational
Sponsor: University of Milan (Other)
Collaborators: International Society of Arthroscopy, Knee Surgery and Orthopaedic Sports Medicine (ISAKOS) (Unknown); ASST Gaetano Pini-CTO (Other)
Responsible Party: Principal Investigator, Pietro Randelli, MD, Prof., MD, University of Milan
Other Study IDs: Lipotendon_LongFu
Record Dates: First submitted 2025-04-16; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Arthroscopic Rotator Cuff Repair; Augmentation; Microfragmented Adipose Tissue
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Treatment group: Cohort of patients that receved a single-row arthroscopic rotator cuff repair, followed by intraoperative injection of autologous microfragmented adipose tissue processed with an enzyme-free technology, 5 years ago in our previous trial (NCT02783352).
  Interventions: Procedure: magnetic resonance imaging (MRI); Other: VAS, SST, ASES, CMS scores, and strength measurements in external rotation and abduction
- Control group: Cohort of patients that received a single-row arthroscopic rotator cuff repair alone, 5 years ago in our previous trial (NCT02783352).
  Interventions: Procedure: magnetic resonance imaging (MRI); Other: VAS, SST, ASES, CMS scores, and strength measurements in external rotation and abduction

INTERVENTIONS:
Procedure: magnetic resonance imaging (MRI) — All enrolled patients will be contacted again at a minimum follow-up of 5 years, and an MRI of the operated shoulder will also be performed.
Other: VAS, SST, ASES, CMS scores, and strength measurements in external rotation and abduction — All enrolled patients will be contacted again at a minimum follow-up of 5 years, and a clinical evaluation will be performed using the following measurements and scores: VAS, SST, ASES, CMS scores, and strength measurements in external rotation and abduction.

SUMMARY:
Specific Aims :

The aim of this prospective randomized controlled single-blind clinical trial was to evaluate the safety and efficacy of autologous microfragmented lipoaspirate tissue in arthroscopic rotator cuff repair.

The primary goal of this study was to test the following hypothesis: an intraoperative injection of autologous microfragmented adipose tissue processed with an enzyme-free technology could improve the clinical outcomes of single-row arthroscopic rotator cuff repair in terms of points in the Constant-Murley score (CMS) collected at least 5 years after surgery.

Background and Significance:

Rotator cuff surgery was initially proposed at the end of the 19th century and evolved then from open to arthroscopic techniques, rising quickly from a minor niche to a fully recognized subspecialty.

To improve clinical and functional results and reduce the retear rate, new fixation techniques and biological solutions to enhance tendon healing are being developed at a fast pace, as shown by the dramatic increase in the number of articles published per year.

Biological solutions to enhance rotator cuff healing include growth factors and platelet-rich plasma, as well as mesenchymal stem cells (MSCs) and their derivatives.

MSCs are believed to enhance tissue healing mainly through stimulation of local cells via paracrine mechanisms and anti-inflammatory and/or immunomodulatory activity, thus creating a suitable microenvironment for tissue repair.

Autologous microfragmented lipoaspirate tissue has been recently introduced in orthopaedics as an easily available source of adipose derived MSCs (ADSCs) to support and accelerate tissue regeneration. Lipoaspirates contain human ADSCs and produce growth factors, such as platelet-derived growth factor, fibroblast growth factor, transforming growth factor beta, and vascular endothelial growth factor, which play important regulatory roles in cellular functions, including adhesion, chemotaxis, proliferation, migration, matrix synthesis, differentiation, and angiogenesis.

Herewith, autologous microfragmented lipoaspirate tissue is expected to optimize the microenvironment for tendon regeneration. Among many approaches, devices relying on nonenzymatic methods and avoiding the use of additives and other additional manipulations (eg, centrifugation) allow one to harvest, process, and obtain autologous microfragmented lipoaspirate tissue directly in the operative theatre under sterile conditions. This permits immediate use in the same surgical intervention without delays owing to the difficulty of an ex vivo cell expansion and the complexity of the current good manufacturing practice requirements for preparing cells for therapeutic use.

Although several animal studies have been published showing promising results for the use of ADSCs in enhancing the healing of rotator cuff tears, minimal evidence describing augmentation of rotator cuff treatment with lipoaspirate.

Preliminary Studies/Progress Report:

This study is a prospective, randomized, double-blind, controlled clinical trial and represents the final follow-up of an our previous study with short follow-up (2 years). The previous study demonstrated that the intraoperative injection of autologous microfragmented adipose tissue is safe and effective in improving short-term clinical and functional results after single-row arthroscopic rotator cuff repair.

Nevertheless, no significant differences emerged between the groups in terms of rerupture rate, complication rate, number of adverse events, and mid-term clinical outcomes.

A previous in vitro study showed that autologous microfragmented adipose tissue significantly increases the proliferation rate of human tendon stem cells without altering their stemness and differentiation capability. Moreover, treated cells increase the expression of VEGF, which is crucial for the neovascularization of the tissue during the healing process.

Research Design and Method:

At least 5 years after surgery, all enrolled patients in the previous study will be call again and will be asked to complete the ASES, SST, and VAS questionnaire and they will undergo a clinical examination, including the CMS and measurement of isometric strength in shoulder forward flexion, abduction, and external rotation. All strength measures will be performed in triplicate with a dynamometer.

During the same assessment day, the patients would be evaluated with MRI of the operated shoulder in order to assess tendon integrity and calculate rerupture rate according to the classification proposed by Sugaya (types IV and V defined as retears). Atrophy of the supraspinatus muscle belly was evaluated according to Warner and fatty degeneration was classified according to Fuchs.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Full-thickness supraspinatus and infraspinatus tendon tears (C1, C2, and C3 according to the SCOI classification)
* Indication for arthroscopic rotator cuff repair
* Informed consent to participate in the study
* Informed consent to participate for the duration of the study

Exclusion Criteria:

* Partial rotator cuff tendon tears (A1, A2, A3, B1, B2, and B3 according to the SCOI classification)
* Massive rotator cuff tear (C4 according to the SCOI classification)
* Subscapularis tendon tear (grade III, IV, or IV according to Lafosse classification)
* Associated anterior, posterior, or multidirectional shoulder instability
* Indication for repair of a SLAP lesion of the biceps anchor
* Grade III or IV muscle atrophy of the supraspinatus and infraspinatus tendons (according to Goutallier or Fuchs classification)
* Intra-articular hyaluronic acid or corticosteroid infiltration within 3 mo from the planned surgical procedure
* Medical comorbidities contraindicating arthroscopic shoulder surgery
* Local (shoulder, abdominal region, gluteal region) or systemic infection, osteomyelitis, or sepsis
* Diabetes mellitus, untreated thyroid disease, chronic kidney disease, rheumatoid arthritis
* Immunodeficiency
* Chronic disorders involving coagulation, platelet aggregation, or severe coagulopathy
* Severe cardiovascular disease
* Stroke or acute cardiovascular event within 6 mo from the planned surgical procedure
* Weight loss for any cause .30 kg in 12 mo or .10 kg in 12 mo without a cause
* Eating disorders or body dysmorphic disorder
* Varices, phlebitis, or scars next to the planned adipose tissue harvesting site
* Alcohol/drug addiction or psychiatric disease compromising compliance with postoperative protocols
* Pregnancy or breastfeeding women
* Informed consent not accepted

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study is a prospective, randomized, double-blind, controlled clinical trial and represents the final follow-up of an our previous study with short follow-up (2 years). At least 5 years after surgery, all enrolled patients in the previous study will be call again and will be asked to complete the ASES, SST, and VAS questionnaire and they will undergo a clinical examination, including the CMS and measurement of isometric strength in shoulder forward flexion, abduction, and external rotation. All strength measures will be performed in triplicate with a dynamometer.
  During the same assessment day, the patients would be evaluated with MRI of the operated shoulder in order to assess tendon integrity and calculate rerupture rate according to the classification proposed by Sugaya (types IV and V defined as retears). Atrophy of the supraspinatus muscle belly was evaluated according to Warner and fatty degeneration was classified according to Fuchs.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-10-11 (Estimated); Study Completion 2026-04-11 (Estimated)

PRIMARY OUTCOMES:
Comparison between the two groups of the incidence of retears at least 5 years after surgery | 5 years
  The primary goal of this study is to evaluate the long-term effecacy of the use of autologous microfragmented adipose tissue in arthroscopic rotator cuff repair, in terms of estimating the incidence of retears at least 5 years after surgery, as assessed by magnetic resonance imaging (MRI).

SECONDARY OUTCOMES:
Comparison of the Constant-Murley score (CMS) between the two groups at least 5 years after surgery. | 5 years
  A secondary objective is to assess the effecacy of microfragmented autologous adipose tissue in arthroscopic repairs of rotator cuff tears in terms of improvement in the postoperative CMS at the 5-year follow-up.
Comparison between the two groups of the difference in the Visual Analogue Scale (VAS) score at least 5 years after surgery. | 5 years
  A secondary objective is to assess the effecacy of microfragmented autologous adipose tissue in arthroscopic repairs of rotator cuff tears in terms of pain reduction of pain, assessed by VAS, at the 5-year follow-up.
Comparison between the two groups of abduction and external rotation strength at least 5 years after surgery. | 5 years
  A secondary objective is to assess the effecacy of microfragmented autologous adipose tissue in arthroscopic repairs of rotator cuff tears in terms of increase in abduction and external rotation strength after surgery at the 5-year follow-up.
Comparison of the ASES (American Shoulder and Elbow Surgeons score) and SST (Simple Shoulder Test) between the two groups at least 5 years after surgery. | 5 years
  A secondary objective is to assess the effecacy of microfragmented autologous adipose tissue in arthroscopic repairs of rotator cuff tears in terms of improvement in the postoperative ASES and SST scores at the 5-year follow-up.
Comparison between the two groups of the progression of supraspinatus fatty degeneration at least 5 years after surgery | 5 years
  A secondary objective is to assess the effecacy of microfragmented autologous adipose tissue in arthroscopic repairs of rotator cuff repair, as assessed by magnetic resonance imaging (MRI) and graded according to the Fuchs classification, at the 5-year follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Gaetano Pini-CTO, Milan, Italy, Italy

REFERENCES:
- [Background] Vigano M, Lugano G, Perucca Orfei C, Menon A, Ragni E, Colombini A, De Luca P, Randelli P, de Girolamo L. Autologous microfragmented adipose tissue reduces inflammatory and catabolic markers in supraspinatus tendon cells derived from patients affected by rotator cuff tears. Int Orthop. 2021 Feb;45(2):419-426. doi: 10.1007/s00264-020-04693-9. Epub 2020 Jul 8. PMID 32642826
- [Background] Fuchs B, Weishaupt D, Zanetti M, Hodler J, Gerber C. Fatty degeneration of the muscles of the rotator cuff: assessment by computed tomography versus magnetic resonance imaging. J Shoulder Elbow Surg. 1999 Nov-Dec;8(6):599-605. doi: 10.1016/s1058-2746(99)90097-6. PMID 10633896
- [Background] Warner JJ, Higgins L, Parsons IM 4th, Dowdy P. Diagnosis and treatment of anterosuperior rotator cuff tears. J Shoulder Elbow Surg. 2001 Jan-Feb;10(1):37-46. doi: 10.1067/mse.2001.112022. PMID 11182734
- [Background] Sugaya H, Maeda K, Matsuki K, Moriishi J. Repair integrity and functional outcome after arthroscopic double-row rotator cuff repair. A prospective outcome study. J Bone Joint Surg Am. 2007 May;89(5):953-60. doi: 10.2106/JBJS.F.00512. PMID 17473131
- [Background] Randelli P, Menon A, Ragone V, Creo P, Bergante S, Randelli F, De Girolamo L, Alfieri Montrasio U, Banfi G, Cabitza P, Tettamanti G, Anastasia L. Lipogems Product Treatment Increases the Proliferation Rate of Human Tendon Stem Cells without Affecting Their Stemness and Differentiation Capability. Stem Cells Int. 2016;2016:4373410. doi: 10.1155/2016/4373410. Epub 2016 Jan 6. PMID 27057170
- [Background] Soleymaninejadian E, Pramanik K, Samadian E. Immunomodulatory properties of mesenchymal stem cells: cytokines and factors. Am J Reprod Immunol. 2012 Jan;67(1):1-8. doi: 10.1111/j.1600-0897.2011.01069.x. Epub 2011 Sep 23. PMID 21951555
- [Background] Shi M, Liu ZW, Wang FS. Immunomodulatory properties and therapeutic application of mesenchymal stem cells. Clin Exp Immunol. 2011 Apr;164(1):1-8. doi: 10.1111/j.1365-2249.2011.04327.x. Epub 2011 Feb 24. PMID 21352202
- [Background] Schmitt A, van Griensven M, Imhoff AB, Buchmann S. Application of stem cells in orthopedics. Stem Cells Int. 2012;2012:394962. doi: 10.1155/2012/394962. Epub 2012 Feb 23. PMID 22550505
- [Background] Mei SH, Haitsma JJ, Dos Santos CC, Deng Y, Lai PF, Slutsky AS, Liles WC, Stewart DJ. Mesenchymal stem cells reduce inflammation while enhancing bacterial clearance and improving survival in sepsis. Am J Respir Crit Care Med. 2010 Oct 15;182(8):1047-57. doi: 10.1164/rccm.201001-0010OC. Epub 2010 Jun 17. PMID 20558630
- [Background] Krasnodembskaya A, Song Y, Fang X, Gupta N, Serikov V, Lee JW, Matthay MA. Antibacterial effect of human mesenchymal stem cells is mediated in part from secretion of the antimicrobial peptide LL-37. Stem Cells. 2010 Dec;28(12):2229-38. doi: 10.1002/stem.544. PMID 20945332
- [Background] Gnecchi M, Zhang Z, Ni A, Dzau VJ. Paracrine mechanisms in adult stem cell signaling and therapy. Circ Res. 2008 Nov 21;103(11):1204-19. doi: 10.1161/CIRCRESAHA.108.176826. PMID 19028920
- [Background] Angeline ME, Rodeo SA. Biologics in the management of rotator cuff surgery. Clin Sports Med. 2012 Oct;31(4):645-63. doi: 10.1016/j.csm.2012.07.003. PMID 23040551
- [Background] Randelli P, Randelli F, Ragone V, Menon A, D'Ambrosi R, Cucchi D, Cabitza P, Banfi G. Regenerative medicine in rotator cuff injuries. Biomed Res Int. 2014;2014:129515. doi: 10.1155/2014/129515. Epub 2014 Aug 13. PMID 25184132
- [Background] McElvany MD, McGoldrick E, Gee AO, Neradilek MB, Matsen FA 3rd. Rotator cuff repair: published evidence on factors associated with repair integrity and clinical outcome. Am J Sports Med. 2015 Feb;43(2):491-500. doi: 10.1177/0363546514529644. Epub 2014 Apr 21. PMID 24753240
- [Background] Randelli P, Cucchi D, Ragone V, de Girolamo L, Cabitza P, Randelli M. History of rotator cuff surgery. Knee Surg Sports Traumatol Arthrosc. 2015 Feb;23(2):344-62. doi: 10.1007/s00167-014-3445-z. Epub 2014 Dec 2. PMID 25448135